CLINICAL TRIAL: NCT05761743
Title: Evaluation of Glycemic Control and Changes in Skeletal Profile in Patients With Type II Diabetes Undergoing Parathyroidectomy for Primary Hyperparathyroidism
Brief Title: Glycemic Control, Type II Diabetes, Parathyroidectomy
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Judy Jin, MD, Physician in Endocrine Surgery, The Cleveland Clinic
Other Study IDs: 22-1407
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Primary Hyperparathyroidism; Type 2 Diabetes
Keywords: Hyperparathyroidism, Glycemic Control
MeSH Terms: conditions — Hyperparathyroidism, Primary; Diabetes Mellitus, Type 2; Hyperparathyroidism | interventions — Urination; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PHPT and DM Patients, Parathyroidectomy: Patients with primary hyperparathyroidism with type 2 diabetes, that decided with their physician/surgeon to continue with a parathyroidectomy (independent of research).
  Interventions: Diagnostic Test: Urine and Blood Test
- PHPT and DM Patients, NO Parathyroidectomy: Patients with primary hyperparathyroidism with type 2 diabetes, that have decided with their physician/surgeon to be managed medically with no parathyroidectomy.
  Interventions: Diagnostic Test: Urine and Blood Test

INTERVENTIONS:
Diagnostic Test: Urine and Blood Test — Urine N-telopeptide and serum osteocalcin

SUMMARY:
The purpose of this study is to assess glycemic control after parathyroidectomy in patients with primary hyperparathyroidism and concomitant type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Primary hyperparathyroidism (PHPT) is known to affect the kidney and skeletal system, however, recent data have suggested that patients can also exhibit an increased cardiovascular risk and metabolic abnormalities Primary hyperparathyroidism (PHPT) is the most common cause of hypercalcemia, with an estimated prevalence of 0.8% in the general population. Type 2 diabetes mellitus (DM) is the most prevalent chronic disease with an estimated prevalence of 10%. Based on the estimated prevalence of this two conditions, we would expect a comorbid prevalence of both diseases in the same individual of approximately 0.08%. However, the prevalence of DM in patients with PHPT is much higher ranging from anywhere 7.8% to 22%, suggesting that this is not mere coincidence.

While the exact mechanism is not clear, in vivo study demonstrated that parathyroid hormone (PTH) reduces the insulin-stimulated uptake as well as decrease glucose transporter and the insulin receptor. Hypercalcemia can also be associated with impaired insulin sensitivity and insufficient suppression of gluconeogenesis. In some patient series, some improvement in glycemic profiles have been shown in patients after parathyroidectomy (PTX).

In addition, both DM and PHPT are known risk factors for the development of bone abnormality patients with DM have increased risk of hip fractures while cortical bone (i.e. the forearm) are more commonly affected in patients with PHPT. There are currently very few studies evaluating the interaction of both conditions in terms of patient skeletal profiles and bone health.

Participants with PHPT and DM will be recruited and followed over the course of a year. There are two groups: the group of patients that decided to pursue a parathyroidectomy, and a group of patients that will be managed non-surgically. Clinical data will be collected along with blood tests.

ELIGIBILITY:
Inclusion Criteria:

1. Study group: Consecutive patients older than 18 years old with concomitant PHPT and DM who will undergo PTX. The indications and need for surgery will be independent from the research team.
2. Control group: Consecutive patients older than 18 years old with concomitant PHPT and DM who will not undergo PTX. The indications to forgo surgery will be independent from the research team.

Exclusion Criteria:

1. Patients with recurrent or persistent PHPT will not be included.
2. Patients who are included but have evidence of recurrent or persistent PHPT based on six-month laboratory workup will be excluded from the final analysis (<5% expected)9.
3. Patients with type 1 diabetes mellitus
4. Patients with secondary and/or tertiary hyperparathyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a multi-specialty academic medical center coming in to see their physician for surgery, and/or management of their PHPT and DM.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Assess glycemic control after parathyroidectomy in patients with primary hyperparathyroidism and concomitant type 2 diabetes mellitus | 1 year
  Preoperative, operative and postoperative variables will be compared between groups using the unpaired T-test and Chi-squared test for continuous and categorical variables, respectively. Postoperative differences compared to the baseline will be analyzed using a paired T-test.

SECONDARY OUTCOMES:
Assess the changes in skeletal profile after parathyroidectomy in patients with primary hyperparathyroidism and concomitant type 2 diabetes mellitus | 1 year
  Preoperative, operative and postoperative variables will be compared between groups using the unpaired T-test and Chi-squared test for continuous and categorical variables, respectively. Postoperative differences compared to the baseline will be analyzed using a paired T-test.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Jin, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No